CLINICAL TRIAL: NCT04670016
Title: Health Related Quality of Life (HRQL) and Symptom Assessment in Patients Diagnosed With Diffuse Intrinsic Pontine Glioma (DIPG) or Recurrent and Re-irradiated Brain Tumours and Their Caregivers: A Non-Therapeutic Study
Brief Title: HRQL and Symptom Assessment for Patients With DIPG or Recurrent and Re-irradiated Brain Tumours and Their Caregivers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: University of Toronto (Other); Université de Montréal (Other); University of Ottawa (Other); Western University, Canada (Other); McMaster University (Other); Alberta Children's Hospital (Other); Stollery Children's Hospital (Other); British Columbia Children's Hospital (Other); CancerCare Manitoba (Other); Children's Hospital of Eastern Ontario (Other); The Hospital for Sick Children (Other); McMaster Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); St. Justine's Hospital (Other); Montreal Children's Hospital of the MUHC (Other); IWK Health Centre (Other); Janeway Children's Health and Rehabilitation Centre (Unknown); Princess Margaret Hospital, Canada (Other); London Health Sciences Centre (Other); The Ottawa Hospital (Other); CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Fiona Simone Maria Schulte, ssistant Professor in the Department of Oncology, Division of Psychosocial Oncology in the Cumming School of Medicine, University of Calgary
Other Study IDs: HREBA.CC-16-0821
Record Dates: First submitted 2020-11-17; First posted 2020-12-17 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: DIPG; Brain Tumor, Pediatric, Recurrent; Brain Tumor, DIPG; Radiation Toxicity; Radiation Exposure; Brain Tumor, Pediatric
Keywords: health-related quality of life; psychosocial; re-irradiation; DIPG; pediatric brain tumor
MeSH Terms: conditions — Brain Neoplasms; Recurrence; Diffuse Intrinsic Pontine Glioma; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient/Caregiver dyad diagnosed with DIPG: All of these criteria must be met for a patient to be eligible for this study:
  1. Patient aged >2 and <21 years treated with a repeat course of radiation for DIPG
  2. Radiation for the first tumour must be a primary brain neoplasm (i.e. not leukemia).
  3. Enrollment within 14 days of starting re-irradiation (RT2).
  4. Patients with malignant transformation of the first tumour are eligible.
  5. There are no restrictions on histology or RT1/RT2 dose-fractionation or RT2 body site. In other words, RT2 may be directed at a different location to RT1.
  6. The patient is treated at a site where the study is approved by the local ethics board
  7. Consent, and, if applicable, assent, has been obtained according to institutional standards
  Interventions: Other: This study does not include an intervention.
- Patient/Caregiver dyad with re-RT for a recurrent brain tumour: All of these criteria must be met for a patient to be eligible for this study:
  1. Patient aged >2 and <21 years treated with a repeat course of radiation for a recurrent or progressive brain tumour (stratum 2).
  2. Radiation for the first tumour must be a primary brain neoplasm (i.e. not leukemia).
  3. Enrollment within 14 days of starting re-irradiation (RT2).
  4. Patients with malignant transformation of the first tumour are eligible.
  5. There are no restrictions on histology or RT1/RT2 dose-fractionation or RT2 body site. In other words, RT2 may be directed at a different location to RT1.
  6. The patient is treated at a site where the study is approved by the local ethics board
  7. Consent, and, if applicable, assent, has been obtained according to institutional standards
  Interventions: Other: This study does not include an intervention.

INTERVENTIONS:
Other: This study does not include an intervention. — This study does not include an intervention.

SUMMARY:
Although many children with brain tumours are successfully cured of their disease, a substantial proportion of patients suffer disease recurrence and require further treatment. This therapy may involve a repeat course of radiation (RT2). Based on retrospective data, re-irradiation may provide palliative and even potentially curative benefit. However, such retrospective data are subject to bias, which may over-report survival and under-report toxicity. Furthermore, we do not know how re-irradiation affects patients' HRQOL. The goal of this research is to prospectively describe the HRQOL of patients diagnosed with DIPG and recurrent brain tumors and their families before and after re-irradiation to more accurately assess the benefit versus the toxicity of this treatment.

In addition, if we are able to demonstrate the feasibility of collecting HRQOL information on a routine basis we will be able to justify the need to conduct this research further and implement HRQOL screening as a standard of care for these patients. Re-irradiation for children with DIPG and recurrent brain tumours will not cure these children from their disease but may improve neurological function and wellbeing. We postulate that the opportunity of more time to say the final good bye and creating memories will facilitate bereavement and prevent psychological dysfunction of parents and siblings. A greater understanding of what helps these families may enable clinicians to better support these children and their families in this difficult disease course. Ultimately our goal is to improve the psychological experience of these patients and their families.

DETAILED DESCRIPTION:
Many children diagnosed with brain tumours are at significant risk of disease recurrence following their initial treatment, with recurrence rates ranging from 30-100% depending on the type of brain tumour. Disease recurrence represents a serious clinical issue in brain tumour patients and when this occurs, additional treatment is needed. These treatments may result in further damage to the surrounding normal brain tissue, resulting in neurocognitive decline (brain or mental function) and reduced quality of life. A novel treatment option for these patients is to administer a second course of radiation (re-irradiation). However, the effects of re-irradiation on quality-of-life are poorly studied. This study aims to increase the knowledge surrounding re-irradiation, particularly with regards to HRQOL.

The primary objective of the proposed study is to describe the HRQOL and symptoms for children diagnosed with DIPG or recurrent brain tumours treated with repeat radiation and their caregivers over time.

We have four Aims. Aim 1: To describe the HRQOL trajectory and symptoms for children diagnosed with DIPG and in children treated with re-irradiation for a recurrent brain tumour and their caregivers over time. Aim 2: To identify critical time points of HRQOL difficulty across the trajectory of DIPG/recurrent brain tumour treatment and to ascertain demographic and/or medical sequelae that are related to HRQOL outcomes. Aim 3: To determine the feasibility of conducting routine assessment of HRQL in children diagnosed with DIPG/recurrent brain tumours and their caregivers based on recruitment and retention rates. Aim 4: To report the incidence of radiation necrosis (RN), local control, progression-free survival and overall survival after re-irradiation.

Our goal to is enroll 25 to 30 patient/caregiver dyads diagnosed with DIPG and 32 patient/caregiver dyads treated with re-RT for a recurrent/progressive brain tumour onto the trial over the study period and to follow patients until their disease progresses again, which has been, on average, 6 months after completion of RT2.

Once deemed eligible, individual patient recruitment will be the responsibility of the institution Clinical Research Assistant (CRA). Upon consenting to take part in the study, patients and families will be contacted using an online administration and scoring program. HRQOL assessments will take 15-25 minutes to complete at each time point. Baseline questionnaires will be completed at the time of recurrence or progressive DIPG or other brain tumor (+/- 7 days from start of treatment, maximum 14 days). Patients will then complete HRQOL measures at the end of re-irradiation and then again every two months.

Necrosis and local tumour control will be assessed using MRI ordered as part of standard-of-care follow-up (recommended scan interval every 3-6 months until 5 years post-treatment). Necrosis and other toxicities, if present without evidence of disease recurrence, will be graded at baseline and each post-RT2 standard-of-care visit using CTCAE v5.0 (a rating scale of side effects). Steroid use and Lansky play score will be recorded at each visit. Progression and death will be collected from the health record. Re-irradiation dosimetry (in electronic RT-DICOM format) will be requested for all enrolled patients.

Study measures will be available in both English and French. HRQOL measures will include: the Pediatric Quality of Life (PedsQL) General module; the PedsQL Brain Tumour module; the PedsQL Family Impact module; and the Short Form 36 (SF-36), to assess parent quality of life via physical and mental health functioning subscales. Children who require help completing questionnaires will be aided by a CRA. For those 2 to 5 years of age or those who have cognitive disability that impairs their ability to self-report as assessed by their parents, proxy-report by parent or caregiver will be used.

The Symptom Screening in Pediatrics Tool (SSPedi) will also be used to screen for pediatric cancer symptoms.

The Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety, Depressive Symptoms, and Pain Interference measures short forms will be administered to screen for current symptoms of anxiety, depression and assess pain interference.

A linear mixed models approach will be used to compare HRQOL outcomes over time. Further, HRQOL outcomes will be compared across assessment time points and paired sample t-tests will be conducted to identify critical periods of significantly lower and/or higher HRQOL for patients and caregivers. Correlational analyses will be used to explore variables that might emerge as related to HRQL outcome scores. Recruitment rates (patients participating vs. patients eligible) and retention rates (non-completion, lost to follow-up) will be examined. Finally, all incident cases of radiation necrosis without obvious tumour progression will be examined, while accounting for competing risks of disease progression and death from any cause.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged >2 and <21 years treated with a repeat course of radiation for DIPG or other recurrent or progressive brain tumour.
2. Radiation for the first tumour must be a primary brain neoplasm (i.e. not leukemia).
3. Enrollment within 14 days of starting re-irradiation (RT2).
4. Patients with malignant transformation of the first tumour are eligible.
5. There are no restrictions on histology or RT1/RT2 dose-fractionation or RT2 body site. In other words, RT2 may be directed at a different location to RT1.
6. The patient is treated at a site where the study is approved by the local ethics board
7. Consent, and, if applicable, assent, has been obtained according to institutional standards

Exclusion Criteria:

1. Inability to complete questionnaires in English or French.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Up to 30 patients diagnosed with DIPG and up to 32 patients diagnosed with another recurrent or progressive brain tumor will be enrolled in this study.
  There will be no registration on study for screening purposes only. Eligible patients who consent to this study therapy will be registered at the PI's institution, specifically with the PI's research coordinator. A study subject number will be assigned to the patient upon registration.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (HRQOL) for children diagnosed with DIPG and in children treated with re-irradiation for a recurrent brain tumour | 2 months after the second radiation
  Health-related quality-of-life will be measured using the Pediatric Quality of Life Inventory (PedsQL) General Core Scales

SECONDARY OUTCOMES:
HRQOL disease specific modules and family impact | 2 months after the second radiation]
  PedsQL Brain Tumor and Family Impact Module
Symptom burden for children diagnosed with DIPG and in children treated with re-irradiation for a recurrent brain tumour | 2 months after the second radiation]
  Symptom Screening in Pediatrics (SSPEDI)
Caregiver HRQOL | 2 months after the second radiation]
  Short Form 36 (SF-36)
Anxiety, Depression and Pain Interference | 2 months after the second radiation]
  Patient Reported Outcomes Measurement Information System (PROMIS): Anxiety, Depression and Pain Interference Short Forms
Radiation necrosis (RN), local control, progression-free survival and overall survival after re-irradiation. | 12 months
  Radiation necrosis without obvious tumour progression

OTHER OUTCOMES:
Feasibility of conducting routine assessment of HRQOL in children diagnosed with DIPG/recurrent brain tumours and their caregivers. | 4 months after the second radiation
  Recruitment (patients participating vs. patients eligible) and retention rates

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Schulte, PhD, Principal Investigator — University of Calgary; Derek Tsang, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (13):
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec

IPD SHARING:
Plan to Share IPD: No